CLINICAL TRIAL: NCT01498653
Title: A Randomised, Double-blind, Double-dummy, Parallel Group Study to Evaluate the Efficacy and Safety of Fluticasone Furoate/Vilanterol Trifenatate (FF/VI) Inhalation Powder Delivered Once Daily Compared to Fluticasone Propionate Delivered Twice Daily in the Treatment of Asthma in Adolescent and Adult Subjects of Asian Ancestry Currently Treated With High-strength Inhaled Corticosteroids or Mid-strength ICS/LABA Combination Therapy.
Brief Title: Evaluating the Efficacy and Safety of Fluticasone Furoate/Vilanterol Trifenatate in the Treatment of Asthma in Adolescent and Adult Subjects of Asian Ancestry
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113714
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/VI 200/25mcg once daily (Experimental): ICS/LABA
  Interventions: Drug: GW685698/GW642444
- Fluticasone propionate 500mcg twice daily (Active Comparator): ICS
  Interventions: Drug: CCI18781

INTERVENTIONS:
Drug: GW685698/GW642444 — ICS/LABA
  Arms: FF/VI 200/25mcg once daily
Drug: CCI18781 — ICS
  Arms: Fluticasone propionate 500mcg twice daily

SUMMARY:
A randomised, double-blind, double-dummy, parallel group study to evaluate the efficacy and safety of fluticasone furoate/vilanterol trifenatate (FF/VI) inhalation powder delivered once daily in the treatment of asthma in adolescent and adult subjects of Asian ancestry currently treated with high-strength inhaled corticosteroids or mid-strength ICS/LABA combination therapy

DETAILED DESCRIPTION:
This will be a randomized, double-blind, active-comparator, parallel group, multi-center study. At Visit 1 (Screening Visit) subjects who meet all of the inclusion criteria and none of the exclusion criteria will enter a two week Run-in period. Subjects will remain on their current ICS therapy throughout the Run-in period. At the end of the Run-in period (Visit 2) subjects meeting the randomization criteria will enter a 12 week treatment period and receive one of the two following treatments: 1) FF (200mcg)/VI (25mcg) administered once daily in the evening via a Novel Dry Powder Inhaler (NDPI) 2) Fluticasone propionate 500mcg administered twice daily via DISKUS™ Inhaler In addition, all subjects will be supplied with albuterol/salbutamol inhalation aerosol to be used as required to treat asthma symptoms.

Subjects who have not met the randomization criteria at Visit 2 will be withdrawn from the study.

Subjects meeting the randomization criteria will be randomized to one of the two treatment groups and will attend the clinic for 3 on-treatment visits at Week 4 (Visit 3), Week 8 (Visit 4) and Week 12 (Visit 5). Subjects will receive treatment for 12 weeks. A Follow-up Visit or Contact (Visit 6) will take place 1 week after completing study medication. All clinic visits will take place in the morning. Subjects will participate in the study for a maximum of 15 weeks (Screening to Follow-up inclusive). A subject is regarded to have completed the study if they complete all phase of the study (Screening, treatment, Follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: All subjects must be able and willing to give written informed consent to take part in the study
2. Type of Subject: Outpatients, of Asian ancestry, 12 years of age or older at Visit 1 (or ≥18 years of age or older if local regulations or the regulatory status of study medication permit enrolment of adults only) with a diagnosis of asthma as defined by the Global Initiative for Asthma [GINA, 2009] at least 12 weeks prior to Visit 1.
3. Gender: Male or Eligible Female, defined as non-childbearing potential or childbearing potential using an acceptable method of birth control consistently and correctly
4. Severity of Disease: A best FEV1 of 40%-90% of the predicted normal value at the Visit 1 Screening visit. Predicted values will be based upon NHANES III using the Asian adjustment
5. Reversibility of Disease: Demonstrated ≥12% and ≥200mL reversibility of FEV1 within 10-40minutes following 2-4 inhalations of albuterol/salbutamol inhalation aerosol (or one nebulized treatment with albuterol/salbutamol solution) at the Screening Visit.
6. Current Anti-Asthma Therapy: All subjects must be using an ICS, with or without LABA, for at least 12 weeks prior to Visit 1.
7. Short-Acting Beta2-Agonists: All subjects must be able to replace their current short-acting beta2-agonists with albuterol/salbutamol inhaler at Visit 1 for use as needed for the duration of the study. Subjects must be able to withhold albuterol/salbutamol for at least 4 hours prior to study visits.

Exclusion Criteria:

1. History of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 10 years.
2. Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 and led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
3. Asthma Exacerbation: Any asthma exacerbation requiring oral corticosteroids within 12 weeks of Visit 1 or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to Visit 1.
4. Concurrent Respiratory Disease: A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.
5. Other Concurrent Diseases/Abnormalities: A subjects must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the patient at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
6. Oropharyngeal Examination: A subject will not be eligible for the Run-in if he/she has clinical visual evidence of candidiasis at Visit 1.
7. Allergies:

   * Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the new powder inhaler
   * Milk Protein Allergy: History of severe milk protein allergy.
8. Concomitant Medications: Use of the protocol defined prohibited medications within the prohibited time intervals prior to Screening (Visit 1) or during the study.
9. Tobacco Use: Current smoker or a smoking history of 10 pack years (e.g., 20 cigarettes/day for 10 years). A subject may not have used inhaled tobacco products within the past 3 months (i.e., cigarettes, cigars, smokeless or pipe tobacco).
10. Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating Investigator, sub Investigator, study coordinator, or employee of the participating Investigator.
11. Previous Participation: A subject may not have previously been randomized to treatment in another Phase III FF/VI combination product study
12. Compliance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, disease, or geographical location which seems likely (in the opinion of the Investigator ) to impair compliance with any aspect of this study protocol, including visit schedule and completion of the daily diaries

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- China (6):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
- Philippines (2):
  - GSK Investigational Site, Lipa City
  - GSK Investigational Site, Quezon City
- South Korea (6):
  - GSK Investigational Site, Bucheon-si, Gyeonggi-Do
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Ilsanseo-gu, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lin J, Kang J, Lee SH, Wang C, Zhou X, Crawford J, Jacques L, Stone S. Fluticasone furoate/vilanterol 200/25 mcg in Asian asthma patients: a randomized trial. Respir Med. 2015 Jan;109(1):44-53. doi: 10.1016/j.rmed.2014.10.012. Epub 2014 Oct 31. PMID 25524507
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113714 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 313 participants were randomized to treatment. However, 4 participants were randomized in error and did not receive any study treatment; thus, these participants were not included in the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received >=1 dose of trial medication.
Pre-assignment Details: At screening, participants who meet all of the inclusion criteria entered a 2-week Run-in period. Participants continued on inhaled corticosteroid (ICS) therapy throughout the Run-in period. At the end of the Run-in period, participants meeting the randomization criteria entered a 12-week Treatment Period and received one of the two treatments.
Groups:
- Fluticasone Furoate/Vilanterol 200/25 µg Once Daily: Participants received fluticasone furoate (FF)/vilanterol (VI) 200/25 micrograms (µg) once daily (OD) in the evening,via a Dry Powder Inhaler (DPI), for a period of 12 weeks.
- Fluticasone Propionate 500 µg Twice Daily (BID): Participants received fluticasone propionate (FP) 500 µg inhalation powder BID (in the morning and evening), via the DISKUS, for a period of 12 weeks.
Period: Overall Study
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Started | 155 | 154
Completed | 136 | 119
Not Completed | 19 | 35
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 12 | 26
Not completed — Protocol Violation | 0 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Furoate/Vilanterol 200/25 µg OD: Participants received fluticasone furoate (FF)/vilanterol (VI) 200/25 micrograms (µg) once daily (OD) in the evening, via a Dry Powder Inhaler (DPI), for a period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg OD | Fluticasone Propionate 500 µg Twice Daily (BID) | Total
Number analyzed (Participants) | 155 | 154 | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (12.93) | 48.8 (13.41) | 47.9 (13.19)
Gender [Count of Participants; unit: Participants]
  Female | 96 | 86 | 182
  Male | 59 | 68 | 127
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - East Asian Heritage | 128 | 127 | 255
  Asian - South East Asian Heritage | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (BL) in Daily Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the 12-week Treatment Period
Description: Peak Expiratory Flow is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline was calculated as the value of the averaged daily PM PEF over the 12-week Treatment Period minus the Baseline value. Analysis was performed using Analysis of Covariance (ANCOVA) with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12 (up to Day 84)
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received >=1 dose of trial medication. The primary endpoint analysis only included participants who had PM PEF data for >=4 days in the BL week prior to randomization and >=4 days after randomization. Only participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Groups:
- Fluticasone Furoate/Vilanterol 200/25 µg Once Daily: Participants received fluticasone furoate (FF)/vilanterol (VI) 200/25 micrograms (µg) once daily (OD) in the evening, via a Dry Powder Inhaler (DPI), for a period of 12 weeks.
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Number analyzed (Participants) | 154 | 152
Liters/minute (L/min) | 39.1 (3.01) | 10.5 (3.03)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Vilanterol 200/25 µg Once Daily vs Fluticasone Propionate 500 µg Twice Daily (BID); Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 28.5, 95% CI 2-sided [20.1 to 36.9]

2. Secondary Outcome: Mean Change From Baseline in Daily Morning (AM) PEF Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline was calculated as the value of the averaged daily AM PEF over the 12-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12 (up to Day 84)
Population: ITT Population. In addition, the analysis only included participants who had PM PEF data for at least 2 days in the Baseline week prior to randomization and at least 2 days after randomization. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Number analyzed (Participants) | 154 | 152
L/min | 46.2 (3.07) | 14.0 (3.10)

3. Secondary Outcome: Mean Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: The number of inhalations of rescue albuterol/salbutamol inhalation aerosol (medication used to relieve symptoms immediately) used during the day and night was recorded by the participants in a daily diary. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered as rescue free. Participants who were rescue free for 24-hour periods during the 12-week Treatment Period were assessed. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline is calculated as the average value during the 12-week Treatment Period minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12 (up to Day 84)
Population: ITT Population. In addition, the analysis only included participants who had rescue-free 24-hour period data for at least 2 days in the Baseline week prior to randomization and at least 2 days after randomization. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Number analyzed (Participants) | 155 | 152
Percentage of rescue-free 24-hr periods | 32.4 (2.95) | 31.5 (2.98)

4. Secondary Outcome: Mean Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: Asthma symptoms were recorded in a daily dairy by the participants every day in the morning and evening before taking any rescue or study medication and before PEF measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered as symptom free. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Participants who were symptom free for 24-hour periods during the 12-week Treatment Period were assessed. Change from Baseline is calculated as the average value during the 12-week Treatment Period minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12 (up to Day 84)
Population: ITT Population. In addition, the analysis only included participants who had symptom-free 24-hour period data for at least 2 days in the Baseline week prior to randomization and at least 2 days after randomization. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Number analyzed (Participants) | 155 | 152
Percentage of symptom-free 24-hr periods | 25.4 (2.74) | 20.6 (2.77)

5. Secondary Outcome: Change From Baseline in Total Asthma Quality of Life Questionnaire (AQLQ) Score at Week 12
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire developed to evaluate the impact of asthma treatments on the quality of life of asthma sufferers. The AQLQ contains 32 items in 4 domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). The 32 items of the questionnaire are averaged to produce one overall quality of life score. The response format consists of a 7-point scale, where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment." Change from Baseline was calculated as the Week 12 value minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Number analyzed (Participants) | 140 | 123
Scores on a scale | 0.80 (0.069) | 0.69 (0.074)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to Study Day 84).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received >=1 dose of trial medication.
Arm/Group | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily | Fluticasone Propionate 500 µg Twice Daily (BID)
Serious Adverse Events (participants affected / at risk) | 1/155 | 2/154
Other Adverse Events (participants affected / at risk) | 23/155 | 26/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily (N=155) | Fluticasone Propionate 500 µg Twice Daily (BID) (N=154)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate/Vilanterol 200/25 µg Once Daily (N=155) | Fluticasone Propionate 500 µg Twice Daily (BID) (N=154)
Upper respiratory tract infection (Infections and infestations) | 13 | 18
Nasopharyngitis (Infections and infestations) | 6 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.